CLINICAL TRIAL: NCT03948984
Title: Assessing the Impact of LIve Music in the Intensive Care Unit (ICU) to Improve Care for Critically Ill Patients: A Pilot, Prospective, Single-center Study of Therapeutic Music
Brief Title: Assessing the Impact of LIve Music in the Intensive Care Unit (ICU) to Improve Care for Critically Ill Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Joseph Schlesinger, Assistant Professor of Anesthesiology, Vanderbilt University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 190812
Record Dates: First submitted 2019-05-06; First posted 2019-05-14 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Anxiety; Pain; Critical Illness; Relaxation
MeSH Terms: conditions — Anxiety Disorders; Pain; Critical Illness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Therapeutic Music Session (Experimental)
  Interventions: Behavioral: Therapeutic Music Session

INTERVENTIONS:
Behavioral: Therapeutic Music Session — The 20 minute therapeutic music session will consist of classical music performed by a pianist with or without flute accompaniment with an individual patient's ICU room.

SUMMARY:
Noise in the ICU can worsen patient outcomes through factors such as increased cardiovascular stress, alteration in sleep, and increased discomfort or pain The purpose of this study is to determine the benefit of therapeutic music in the ICU on patients, their families, and ICU staff.

DETAILED DESCRIPTION:
Noise in the ICU can worsen patient outcomes through factors such as increased cardiovascular stress, alteration in sleep, and increased discomfort or pain. The purpose of this study is to determine the benefit of therapeutic music in the ICU on patients, their families, and ICU staff. The results of this study will inform clinicians on best practices for redesigning, implementing and evaluating a patient and family focused therapeutic music program in the ICU.

ELIGIBILITY:
Patient Inclusion Criteria:

* Current hospitalization in adult ICU at Vanderbilt University Medical Center

Patient Exclusion Criteria:

* Airborne or special contact isolation
* Unstable hypotension or bradycardia
* Pregnancy
* Current prisoner status
* The inability to communicate either verbally or in writing in English to complete the therapeutic music evaluations
* Refusal to participate

Family Member Inclusion Criteria

* Family member of ICU patient

Family Member Exclusion Criteria

* The inability to communicate either verbally or in writing English to complete the therapeutic music evaluations
* Refusal to participate

ICU Clinical Staff Inclusion Criteria

* ICU clinical staff who are in the patient's room during the music session

ICU Clinical Staff Exclusion Criteria

* Refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2022-05-31 (Actual); Primary Completion 2025-02-02 (Actual); Study Completion 2025-02-02 (Actual)

PRIMARY OUTCOMES:
Change in perceived pain visual analog score | Immediately before and after therapeutic music session (about 20 minutes long)
  Comparison of patient reported perceived pain visual analog score using an 11-point numerical rating scale ranging from 0 (no pain) to 10 (worst possible pain).
Change in perceived anxiety visual analog score | Immediately before and after therapeutic music session (about 20 minutes long)
  Comparison of patient reported perceived anxiety visual analog score using an 11-point numerical rating scale ranging from 0 (no anxiety) to 10 (worst possible anxiety).
Change in perceived relaxation visual analog scale | Immediately before and after therapeutic music session (about 20 minutes long)
  Comparison of patient reported perceived relaxation visual analog score using an 11-point numerical rating scale ranging from 0 (not relaxed at all) to 10 (completely relaxed).

SECONDARY OUTCOMES:
Acceptability of Intervention Measure (AIM) | After conclusion of therapeutic music session (about 20 minutes)
  Assessment of acceptability of therapeutic music session using the AIM which is a 4-item survey where each item is scored on a 5-point Likert scale ranging from 1 (completely disagree) to 5 (completely agree). Higher total AIM scores indicate greater implementability. This assessment will be completed by patients, family members, and ICU clinical staff.
Patient Perceived Impact | After conclusion of therapeutic music session (about 20 minutes)
  Patient and family member perceived impact will be assessed using the Patient Music Evaluation Form. Patient and family member participants will complete this 2-item word choice question form to assess how live music made them feel (26 word choices offered eg., happy, sad, hopeful, energized) and whether the music performance made them do anything (20 word choices offered eg., laugh, smile, sing).
Feasibility of Intervention (FIM) | After conclusion of therapeutic music session (about 20 minutes)
  ICU clinical staff perceived feasibility of therapeutic music session intervention will be assessed with the FIM, a 4-item, 5-point Likert scale ranging from 1 (completely disagree) to 5 (completely agree). Higher total scores indicate greater feasibility.
Intervention Appropriateness Measure (IAM) | After conclusion of therapeutic music session (about 20 minutes)
  Assessment of appropriateness of therapeutic music session using the IAM which is a 4-item survey where each item is scored on a 5-point Likert scale ranging from 1 (completely disagree) to 5 (completely agree). Higher total AIM scores indicate greater implementability. This assessment will be completed by ICU clinical staff.
Perceived Barriers | After conclusion of therapeutic music session (about 20 minutes)
  Perceived barriers will be assessed using qualitative analysis of a 2-item multiple response option and open-ended questions asking for feedback about facilitation and barriers to implementation of therapeutic music in ICU.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph J. Schlesinger, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No